CLINICAL TRIAL: NCT00193102
Title: Phase II Study of Thalidomide in Combination With Capecitabine in Patients With Metastatic Breast Cancer
Brief Title: Thalidomide in Combination With Capecitabine in Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 60
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Thalidomide; Capecitabine

INTERVENTIONS:
Drug: Thalidomide — Thalidomide
Drug: Capecitabine — Capecitabine

SUMMARY:
The lack of non-overlapping toxicities between the two drugs, the ease of all oral drug administration, and the possibility for antitumor synergy make exploration of this combination regimen attractive in women with previously treated metastatic breast cancer. This phase II trial will be performed in collaboration with the Minnie Pearl Cancer Research Network, a multicenter, community-based clinical trials group.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

Thalidomide + Capecitebine

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic breast cancer confirmed by biopsy
* Measurable or evaluable disease
* Females > 18 years
* Able to perform activities of daily living with minimal assistance
* Life expectancy > 3 months
* Adequate bone marrow, liver and kidney function
* All patients must give written informed consent in order to participate.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Women who are pregnant or lactating.
* Received more than 3 prior chemotherapy regimens in the metastatic setting.
* Received continuous infusion 5-fluorouracil lasting > 120 hours.
* Received thalidomide or capecitabine as their last prior regimen.
* Preexisting moderate to severe neuropathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-04; Primary Completion 2005-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Burris HA 3rd, Jones SF, Shipley D, Meluch AA, Greco FA, Barton JH, Yardley DA, Hainsworth JD. Phase II study of capecitabine in combination with thalidomide in patients with metastatic breast cancer. Cancer Invest. 2010 May;28(4):408-12. doi: 10.3109/07357901003631049. PMID 20210519